CLINICAL TRIAL: NCT05029960
Title: Tolerability and Activity of Brivaracetam (BRV) in Patients With Diffuse Gliomas
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Thomas Wychowski, Associate Professor - Department of Neurology , Epilepsy (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBRT21074
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Brivaracetam; Epilepsy
MeSH Terms: conditions — Brain Neoplasms; Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Brivaracetam at a dose of 50 mg twice daily for 6 months
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Dose of 50 mg twice daily for 6 months

SUMMARY:
The purpose of this study is to determine whether the study medication, brivaracetam, is tolerable and safe for patients with brain tumors.

DETAILED DESCRIPTION:
In this study, subjects will receive usual treatment for their brain tumor. In addition, they will be given brivaracetam at a dose of 50 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with pathologic diagnosis of a supratentorial diffuse astrocytic or oligodendroglial tumor
* Patients must be able to provide informed consent

Exclusion Criteria:

* A pre-existing seizure disorder or epilepsy syndrome prior to tumor diagnosis
* Active maintenance therapy with an antiepileptic seizure drug (AED) prior to diagnosis of tumor
* Patients who have experienced an epileptic seizure as the presenting symptom of their brain tumor
* Predicted life expectancy of less than 6 months from the time of screening
* Pregnancy
* Patients with clinically significant hepatic disease (elevated aminotransferases [bilirubin, alkaline phosphatase] > 3 times upper limit normal)
* Patients with stage 4 or greater renal disease (GFR <30 mL/min/1.73 m2)
* Patients who are unable to swallow a tablet
* Patients with active suicidal ideation or a history of suicide attempt or other serious psychiatric disorder having required hospitalization within the previous 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Brivaracetam | 6 Months
  Evaluate adverse events

SECONDARY OUTCOMES:
Voluntariness for study participation | 6 Months
  Number of people that declined to participate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided